CLINICAL TRIAL: NCT06839417
Title: Effect of Squash Exercise Intervention on Sleep and Mental Health Among Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Yanwei You, Postdoctoral Researcher, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024THZWYY05
Record Dates: First submitted 2025-02-09; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Sleep; Mental Health; Exercise
Keywords: sleep; exercsie; squash
MeSH Terms: conditions — Psychological Well-Being; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise (Experimental): two group two test
  Interventions: Behavioral: Exercise
- control (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — using squash exercise
  Arms: exercise

SUMMARY:
Dear Squash Enthusiast, Hello!

First of all, thank you for participating in this survey! This questionnaire is part of a joint study conducted by the Sports and Brain Science Research Team at Tsinghua University and the Squash program students from Nanjing Sport Institute. The study focuses on promoting squash, understanding the exercise experiences of squash participants, and examining the effects of squash on sleep and mental health. Completing the questionnaire will take approximately 5 minutes.

This research strictly follows the guidelines of the Tsinghua University Ethics Review Committee. All tests are harmless to the body, and there are no right or wrong answers to the questions in the survey. Please respond according to your personal situation. Your personal information will only be used for statistical purposes, and we will ensure that your information is kept strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* (1) healthy young adults ; (2) without chronic diseases or psychiatric disorders between the ages of 18 and 35; (3) absence of regular exercise for the past half year; (4) right-handedness; (5) Neither color blindness nor color weakness exist.

Exclusion Criteria:

* the exclusion criteria includes individuals with a history of cardiovascular, metabolic, or neurological disorders (such as hypertension, diabetes, epilepsy, or other significant medical conditions), as well as those with current or past psychiatric disorders, including depression, anxiety, schizophrenia, or other mood or behavioral disorders. Participants who have engaged in regular physical exercise or athletic training within the past six months will also be excluded, as their activity levels may interfere with the results. Left-handed individuals will be excluded, as handedness can affect motor performance and brain activity patterns. Additionally, individuals with any visual impairment affecting color perception, such as color blindness or color weakness, will be excluded. Those currently using medications that affect cognitive function, mood, or physical performance (e.g., antidepressants, anxiolytics, or beta-blockers) will also be excluded, as will individuals with a history of substance abuse or current substance use. Participants with sleep disorders, such as insomnia or sleep apnea, will be excluded to avoid confounding sleep-related outcomes. Lastly, pregnant or breastfeeding individuals, as well as those currently participating in other clinical trials or studies that could interfere with this research, will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
sleep quality | 3 MONTH
  PSQI

SECONDARY OUTCOMES:
mental health | 3 MONTH
  PHQ9

CONTACTS AND LOCATIONS:
Locations (1):
- Tsinghua, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
This study aims to investigate the effects of squash exercise intervention on sleep and mental health. The research will be conducted in two phases. First, we will conduct a cross-sectional survey to assess the baseline relationship between squash participation and sleep quality, as well as mental well-being. Following this, a randomized controlled trial will be implemented, starting with a one-time intervention to observe immediate effects of squash exercise on sleep and mental health. Subsequently, a 10-week intervention will be conducted, with three sessions per week, each lasting one hour, to explore the long-term impact of regular squash exercise on these outcomes. The goal is to provide insights into how squash as a form of physical activity can influence sleep patterns and mental health.
Supporting Information: Study Protocol
Time Frame: From 2025 March to 2027 March